CLINICAL TRIAL: NCT06144762
Title: Precision Imaging for Early Detection and Targeted Treatment Monitoring in Pancreatic Cancer
Acronym: PANC-O-MICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2023-03 PAN
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pancreas Cancer
Keywords: Radiomics; Ovarian cancer; Genomics; Proteomics; Immune Tumor Microenvironment
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms | interventions — Biological Products; Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample and tissue sample (Experimental): Blood sample and tissue sample
  Interventions: Biological: Biological/Vaccine: Blood sample and tissue sample

INTERVENTIONS:
Biological: Biological/Vaccine: Blood sample and tissue sample — During the surgery :
  Tissus sample : primary tumor and metastasis blood sample : 3 EDTA tubes ex vivo MRI data

SUMMARY:
Specifically, in this project, the objective will be developped a model to capture imaging-based tumor heterogeneity with multiscale radiomics approach by obtaining the mirror tumor image at in vivo MRI, ex vivo MRI at histology. This imaging model giving a perfect virtual histology tumor representation will be secondary implemented on routine in vivo clinical MRI for early cancer detection and treatment monitoring. Successful completion of this proposal will lead to a comprehensive non invasive characterisation of pancreatic cancer and will be a game changer in patient management.

DETAILED DESCRIPTION:
With a five-year survival rate of only 3% for the majority of patients, pancreatic cancer is a global healthcare challenge. By the time of diagnosis over half of pancreatic cancers are metastasized. The dire disease situation reflects our inability to diagnose pancreatic cancer early and to effectively treat it. Our failure to diagnose the disease early results in part from the inaccessibility of the organ, difficulties in detecting small pancreatic lesions by conventional imaging approaches, and a poor understanding of the spectrum of heterogeneity in pancreatic cancer. Single time point, single site biopsies cannot assess entire tumor while multiple biopsies at several time points are not feasible in clinical routine. Limitations of invasive sampling may be addressed with non-invasive imaging that captures morphologic and functional information about the entire tumor in space and, if repeated, in time. Radiomics has the potential for "whole tumour virtual sampling" using a single or serial non-invasive examinations in place of biopsies. By approaching images as data able to be mined, instead of merely pictures in conventional radiology, quantitative imaging allows for further information to be extracted from medical images as well as for global assessments across large patient populations. Therefore, these new quantitative approaches hold the promise of detecting pancreatic cancer characteristics that the naked eye alone cannot perceive from conventional medical imaging, opening new doors for personalized medicine in pancreatic cancer. To date, no study has evaluated the value of radiomics at macroscopic (in vivo 1.5T/3TMRI) and microscopic (ex vivo 9.4TMRI) scale for early cancer detection and targeted treatment monitoring. Specifically, in this project, the objective will be developpe a model to capture imaging-based tumor heterogeneity with multiscale radiomics approach by obtaining the mirror tumor image at in vivo MRI, ex vivo MRI at histology. This imaging model giving a perfect virtual histology tumor representation will be secondary implemented on routine in vivo clinical MRI for early cancer detection and treatment monitoring. Successful completion of this proposal will lead to a comprehensive non invasive characterisation of pancreatic cancer and will be a game changer in patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged >18 2.
* Pathologically proven pancreatic cancer which can beneficiate of upfront surgery or delayed surgery followed by neoadjuvant chemotherapy.
* Negative pregnancy test for women of childbearing potential
* Patients affiliated to a social protection system
* Written informed consent signed before project onset.

Exclusion Criteria:

* presence of metastases,
* Patient who will not have surgery
* Pregnant or breastfeeding women
* Mental or psychological state, physical or legal incapacity preventing participation in the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
the integration of in vivo and ex vivo MRI with histology and molecular caracteristic in order to increase the pancreatic cancer detection and therapeutic response monitoring | The day of the surgery
  The diagnostic performance of the radiomic and multiomic algorithm in pancreatic cancer detection and therapeutic response monitoring.

SECONDARY OUTCOMES:
the imaging phenotype of tumor heterogeneity with a multi-scale radiomic approach by obtaining the image mirror tumor at the in vivo scale | The day of the surgery
  Correlation between radiomic maps and pathogenic maps of heterogeneity,
tumor heterogeneity in artificial intelligence-based imaging reflects and can predict underlying histology (proportion of tumor stroma and density of tumor-infiltrating lymphocytes) (tumor detection and response) and genomics, | The day of the surgery
  Correlation between radiomic algorithms and i/underlying histology (proportion of tumor stroma and density of tumor-infiltrating lymphocytes) (tumor detection and response) ii/ genomics
the heterogeneity of tumor biology via non-invasive imaging of different portions of the tumor, | The day of the surgery
  Correlation between radiomic maps and tumour biology (CYTOF, proteomics and transcriptomics),
Correlate MRI results with hematological molecular biology results. | The day of the surgery
  Correlation between radiomic algorithms for tumor detection and cDNA assay

CONTACTS AND LOCATIONS:
Overall Officials: NOUGARET Stephanie, Study Director — INSTITUT REGIONAL DU CANCER DE MONTPELLIER Cancer de Montpellier
Locations (1):
- NOUGARET Stephanie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nougaret S, Lakhman Y, Gourgou S, Kubik-Huch R, Derchi L, Sala E, Forstner R; European Society of Radiology (ESR) and the European Society of Urogenital Radiology (ESUR). MRI in female pelvis: an ESUR/ESR survey. Insights Imaging. 2022 Mar 28;13(1):60. doi: 10.1186/s13244-021-01152-w. PMID 35347481
- [Background] Soyer P, Revel MP, Dohan A, Vernhet-Kovacsik H, Nougaret S, Hoeffel C. Gender diversity in authorship in Diagnostic & Interventional Imaging: Where are we now? Diagn Interv Imaging. 2022 May;103(5):237-239. doi: 10.1016/j.diii.2022.02.001. Epub 2022 Feb 17. No abstract available. PMID 35183485
- [Background] Tardieu M, Lakhman Y, Khellaf L, Cardoso M, Sgarbura O, Colombo PE, Crispin-Ortuzar M, Sala E, Goze-Bac C, Nougaret S. Assessing Histology Structures by Ex Vivo MR Microscopy and Exploring the Link Between MRM-Derived Radiomic Features and Histopathology in Ovarian Cancer. Front Oncol. 2022 Jan 19;11:771848. doi: 10.3389/fonc.2021.771848. eCollection 2021. PMID 35127479
- [Background] Sadowski EA, Thomassin-Naggara I, Rockall A, Maturen KE, Forstner R, Jha P, Nougaret S, Siegelman ES, Reinhold C. O-RADS MRI Risk Stratification System: Guide for Assessing Adnexal Lesions from the ACR O-RADS Committee. Radiology. 2022 Apr;303(1):35-47. doi: 10.1148/radiol.204371. Epub 2022 Jan 18. PMID 35040672
- [Background] Shinagare AB, Sadowski EA, Park H, Brook OR, Forstner R, Wallace SK, Horowitz JM, Horowitz N, Javitt M, Jha P, Kido A, Lakhman Y, Lee SI, Manganaro L, Maturen KE, Nougaret S, Poder L, Rauch GM, Reinhold C, Sala E, Thomassin-Naggara I, Vargas HA, Venkatesan A, Nikolic O, Rockall AG. Ovarian cancer reporting lexicon for computed tomography (CT) and magnetic resonance (MR) imaging developed by the SAR Uterine and Ovarian Cancer Disease-Focused Panel and the ESUR Female Pelvic Imaging Working Group. Eur Radiol. 2022 May;32(5):3220-3235. doi: 10.1007/s00330-021-08390-y. Epub 2021 Nov 30. PMID 34846566
- [Background] Tibermacine H, Rouanet P, Sbarra M, Forghani R, Reinhold C, Nougaret S; GRECCAR Study Group. Radiomics modelling in rectal cancer to predict disease-free survival: evaluation of different approaches. Br J Surg. 2021 Oct 23;108(10):1243-1250. doi: 10.1093/bjs/znab191. PMID 34423347
- [Background] Nougaret S, Vargas HA, Sala E. BJR female genitourinary oncology special feature: introductory editorial. Br J Radiol. 2021 Sep 1;94(1125):20219003. doi: 10.1259/bjr.20219003. No abstract available. PMID 34415200
- [Background] Rouanet P, Rullier E, Lelong B, Maingon P, Tuech JJ, Pezet D, Castan F, Nougaret S; GRECCAR Study Group*. Tailored Strategy for Locally Advanced Rectal Carcinoma (GRECCAR 4): Long-term Results From a Multicenter, Randomized, Open-Label, Phase II Trial. Dis Colon Rectum. 2022 Aug 1;65(8):986-995. doi: 10.1097/DCR.0000000000002153. Epub 2022 Jul 5. PMID 34759247
- [Background] Nougaret S, Tibermacine H, Tardieu M, Sala E. Radiomics: an Introductory Guide to What It May Foretell. Curr Oncol Rep. 2019 Jun 25;21(8):70. doi: 10.1007/s11912-019-0815-1. PMID 31240403
- [Background] Weigelt B, Vargas HA, Selenica P, Geyer FC, Mazaheri Y, Blecua P, Conlon N, Hoang LN, Jungbluth AA, Snyder A, Ng CKY, Papanastasiou AD, Sosa RE, Soslow RA, Chi DS, Gardner GJ, Shen R, Reis-Filho JS, Sala E. Radiogenomics Analysis of Intratumor Heterogeneity in a Patient With High-Grade Serous Ovarian Cancer. JCO Precis Oncol. 2019 Jun 6;3:PO.18.00410. doi: 10.1200/PO.18.00410. eCollection 2019. No abstract available. PMID 32914032
- [Background] Dextraze K, Saha A, Kim D, Narang S, Lehrer M, Rao A, Narang S, Rao D, Ahmed S, Madhugiri V, Fuller CD, Kim MM, Krishnan S, Rao G, Rao A. Spatial habitats from multiparametric MR imaging are associated with signaling pathway activities and survival in glioblastoma. Oncotarget. 2017 Dec 5;8(68):112992-113001. doi: 10.18632/oncotarget.22947. eCollection 2017 Dec 22. PMID 29348883
- [Background] Chu LC, Park S, Kawamoto S, Fouladi DF, Shayesteh S, Zinreich ES, Graves JS, Horton KM, Hruban RH, Yuille AL, Kinzler KW, Vogelstein B, Fishman EK. Utility of CT Radiomics Features in Differentiation of Pancreatic Ductal Adenocarcinoma From Normal Pancreatic Tissue. AJR Am J Roentgenol. 2019 Aug;213(2):349-357. doi: 10.2214/AJR.18.20901. Epub 2019 Apr 23. PMID 31012758
- [Background] Zhang Z, Li S, Wang Z, Lu Y. A Novel and Efficient Tumor Detection Framework for Pancreatic Cancer via CT Images. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:1160-1164. doi: 10.1109/EMBC44109.2020.9176172. PMID 33018193
- [Background] Chu LC, Park S, Kawamoto S, Wang Y, Zhou Y, Shen W, Zhu Z, Xia Y, Xie L, Liu F, Yu Q, Fouladi DF, Shayesteh S, Zinreich E, Graves JS, Horton KM, Yuille AL, Hruban RH, Kinzler KW, Vogelstein B, Fishman EK. Application of Deep Learning to Pancreatic Cancer Detection: Lessons Learned From Our Initial Experience. J Am Coll Radiol. 2019 Sep;16(9 Pt B):1338-1342. doi: 10.1016/j.jacr.2019.05.034. No abstract available. PMID 31492412
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Himoto Y, Veeraraghavan H, Zheng J, Zamarin D, Snyder A, Capanu M, Nougaret S, Vargas HA, Shitano F, Callahan M, Wang W, Sala E, Lakhman Y. Computed Tomography-Derived Radiomic Metrics Can Identify Responders to Immunotherapy in Ovarian Cancer. JCO Precis Oncol. 2019 Aug 15;3:PO.19.00038. doi: 10.1200/PO.19.00038. eCollection 2019. PMID 32914033
- [Background] Meier A, Veeraraghavan H, Nougaret S, Lakhman Y, Sosa R, Soslow RA, Sutton EJ, Hricak H, Sala E, Vargas HA. Association between CT-texture-derived tumor heterogeneity, outcomes, and BRCA mutation status in patients with high-grade serous ovarian cancer. Abdom Radiol (NY). 2019 Jun;44(6):2040-2047. doi: 10.1007/s00261-018-1840-5. PMID 30474722
- [Background] Vargas HA, Veeraraghavan H, Micco M, Nougaret S, Lakhman Y, Meier AA, Sosa R, Soslow RA, Levine DA, Weigelt B, Aghajanian C, Hricak H, Deasy J, Snyder A, Sala E. A novel representation of inter-site tumour heterogeneity from pre-treatment computed tomography textures classifies ovarian cancers by clinical outcome. Eur Radiol. 2017 Sep;27(9):3991-4001. doi: 10.1007/s00330-017-4779-y. Epub 2017 Mar 13. PMID 28289945